CLINICAL TRIAL: NCT05342493
Title: AJOVY Subcutaneous Injection Long-term Specified Use-results Survey
Brief Title: Specified Drug Use Survey on AJOVY Subcutaneous Injection for Long-term Use
Status: Recruiting | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 406-101-00013
Record Dates: First submitted 2022-04-17; First posted 2022-04-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Drug: Ajovy syringe for SC injection 225 mg.
  Interventions: Drug: Fremanezumab 225 Mg/1.5 mL Subcutaneous Solution

INTERVENTIONS:
Drug: Fremanezumab 225 Mg/1.5 mL Subcutaneous Solution — The usual adult dose is 225 mg of fremanezumab (genetical recombination) administered subcutaneously as a single dose once every 4 weeks or 675 mg administered subcutaneously as a single dose once every 12 weeks.

SUMMARY:
To evaluate the long-term safety of AJOVY in patients under actual use conditions and to specifically evaluate cardiovascular events. In addition, information on efficacy will be collected.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* patients with a known hypersensitivity to components of AJOVY

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Japan who are planned to be newly started on Ajovy syringe for SC injection 225 mg therapy for the suppression of migraine attacks
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2029-06-22 (Estimated)

PRIMARY OUTCOMES:
Safety information (Adverse Event) | 2 years from the start date of treatment
  Any untoward medicinal occurrence in a patient or clinical study subject administered a Medicinal Product and which does not necessarily have a causal relationship with this treatment (see Annex Ⅳ, ICH-E2A Guideline).
  An Adverse Event can therefore be any unfavorable and unintended sign (e.g. abnormal laboratory finding), symptom, or disease temporally associated with the use of a Medicinal Product, whether or not it is considered causally related to the Medicinal Product.
Number of Special Situations | 2 years from the start date of treatment
  Collecting any Situations related to the use of an Otsuka product which may or may not be associated with an adverse event:
  * Maternal (pregnancy and breastfeeding) or paternal (via semen) exposure;
  * Exposure during breastfeeding;
  * Overdose/Incorrect dosage, misuse, abuse (e.g. patient sharing products);
  * Medication errors (e.g. patient took wrong dose);
  * Lack of therapeutic efficacy (e.g. the product doesn't work);
  * Occupational exposure (e.g.: nurse administering the product is exposed);
  * Cases of suspected transmission of infectious agents;
  * Use of suspected or confirmed falsified product(s) or quality defect of the product(s);
  * Withdrawal reactions;
  * Accidental exposure (e.g.: child takes parent's product);
  * Drug-drug/drug-food interactions;
  * Unintentional use of product in a non-approved population (e.g.: pediatric or geriatric population);
  * Disease progression/exacerbation of existing disease
Number of off-Label Use | 2 years from the start date of treatment
  Collecting any type of off-Label Use that refers to situations where a product is intentionally used for a medical purpose not in accordance with the authorized product information. Off-label use also includes the intentional use in non-authorized population categories not indicated in the label.
Incidence of Serious Adverse Event (e.g. resulting in death or life-threatening) | 2 years from the start date of treatment
  Collecting the number of any adverse drug experience/event occurring at any dose which
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or prolonged of existing hospitalization
  * results in persistent or significant disability or incapacity
  * is a congenital anomaly/birth defect
  * is medically significant.
Incidence of Non-serious Adverse Events (i.e. all Adverse Events that do not meet the definition of a serious Adverse Event) | 2 years from the start date of treatment
  Collecting the number of non-serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yasuhiko Fukuta, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Pharmacovigilance Department, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No